CLINICAL TRIAL: NCT06038279
Title: A Randomised, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Trial of INI-2004 in Healthy Volunteers and Participants With Allergic Rhinitis.
Brief Title: Trial of INI-2004 in Healthy Volunteers and Participants With Allergic Rhinitis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inimmune Corporation (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INI-2004-101
Record Dates: First submitted 2023-07-31; First posted 2023-09-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2023-09

CONDITIONS: Allergic Rhinitis Due to Weed Pollen; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: This is a Phase I/Ib, randomised, double-blind, placebo-controlled study of INI-2004, administered as single or multiple doses.This study will be conducted in two parts: Phase I (SAD) and Phase Ib (MAD).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study. Blinding of active/placebo assignment is critical to the integrity of this clinical study. Those blinded to study drug assignment include the Sponsor, the PI (or delegate), clinical study personnel participating in participants' care or clinical evaluations, the CRO project team (with exceptions noted below) and the study participants. INI-2004 and placebo will be administered to the participant in a manner to ensure treatment assignment remains blinded. Blinded data will be provided to the SRC so as not to reveal treatment assignment.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Arm 1 (SAD)- INI-2004 Dose Cohort 1 (Experimental): Healthy Participants will be enrolled and randomised to receive a single dose of INI-2004 or placebo intranasally (ratio 3:1 active: placebo).
  Interventions: Drug: INI-2004
- Arm 2 (SAD)- INI-2004 Dose Cohort 2 (Experimental): Healthy Participants will be enrolled and randomised to receive a single dose of INI-2004 or placebo intranasally (ratio 3:1 active: placebo).
  Interventions: Drug: INI-2004
- Arm 3 (SAD)- INI-2004 Dose Cohort 3 (Experimental): Healthy Participants will be enrolled and randomised to receive a single dose of INI-2004 or placebo intranasally (ratio 3:1 active: placebo).
  Interventions: Drug: INI-2004
- Arm 4 (SAD)- INI-2004 Dose Cohort 4 (Experimental): Healthy Participants will be enrolled and randomised to receive a single dose of INI-2004 or placebo intranasally (ratio 3:1 active: placebo).
  Interventions: Drug: INI-2004
- Placebo (Placebo Comparator): Healthy Participants will be enrolled and randomised to receive a single dose of INI-2004 or placebo intranasally (ratio 3:1 active: placebo).
  Interventions: Drug: Placebo
- Arm 1 (MAD) - INI-2004 Dose Cohort 1 (Experimental): Participants with allergic rhinitis will be enrolled and randomised (ratio 3:1 active:placebo) to receive INI-2004 or placebo intranasally once per week for a total of 4 weeks.
  Interventions: Drug: INI-2004
- Arm 2 (MAD) -INI-2004 Dose Cohort 2 (Experimental): Participants with allergic rhinitis will be enrolled and randomised (ratio 3:1 active:placebo) to receive INI-2004 or placebo intranasally once per week for a total of 4 weeks.
  Interventions: Drug: INI-2004
- Arm 3 (MAD) - INI-2004 Dose Cohort 3 (Experimental): Participants with allergic rhinitis will be enrolled and randomised (ratio 3:1 active:placebo) to receive INI-2004 or placebo intranasally once per week for a total of 4 weeks.
  Interventions: Drug: INI-2004
- Placebo (MAD) (Placebo Comparator): Participants with allergic rhinitis will be enrolled and randomised (ratio 3:1 active:placebo) to receive INI-2004 or placebo intranasally once per week for a total of 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INI-2004 — INI-2004 (a toll-like receptor [TLR]4 agonist) liposomal formulation. INI-2004 is an intranasal (IN) TLR4 agonist that is targeted to prevent AR symptoms in subjects with seasonal AR.
  Arms: Arm 1 (MAD) - INI-2004 Dose Cohort 1; Arm 1 (SAD)- INI-2004 Dose Cohort 1; Arm 2 (MAD) -INI-2004 Dose Cohort 2; Arm 2 (SAD)- INI-2004 Dose Cohort 2; Arm 3 (MAD) - INI-2004 Dose Cohort 3; Arm 3 (SAD)- INI-2004 Dose Cohort 3; Arm 4 (SAD)- INI-2004 Dose Cohort 4
Drug: Placebo — The Placebo for INI-2004 is a clear, colorless solution free of particles supplied in 10 mL glass vials with a 10 mL fill.
  Other Names: Placebo for INI-2004
  Arms: Placebo; Placebo (MAD)

SUMMARY:
This is a Phase I/Ib, randomised, double-blind, placebo-controlled study of INI-2004, administered as single or multiple doses. This study will be conducted in two parts: Phase I single ascending dose (SAD) and Phase Ib multiple ascending dose (MAD).

DETAILED DESCRIPTION:
This is a Phase I/Ib, randomised, double-blind, placebo-controlled study of INI-2004, administered as single or multiple doses.

Phase I (SAD) - Healthy Participants will be enrolled and randomised to 4 dose cohorts (n=8 per cohort) to receive single ascending doses of INI-2004 or placebo (ratio 3:1 active: placebo). Dosing in each cohort will commence with two sentinels, with one of the two sentinels randomised to receive INI-2004 and the other randomised to receive placebo. The safety and tolerability of each sentinel participant will be monitored in the clinic until Day 2 and will be reviewed by the Principal Investigator (PI) prior to dosing the remainder of participants in each cohort. The decision to escalate between cohorts will be made by a safety review committee (SRC) following completion of the Day 3 visit for at least 6 out of 8 participants in the cohort. Cohorts will be dosed in an escalating order.

Phase Ib (MAD) - Phase Ib (MAD) may commence following completion of SAD Cohort 3 or SAD Cohort 4.

Up to 3 dose levels are planned to be evaluated. To be eligible for study inclusion, participants must have a positive response to the ragweed nasal allergen challenge at screening. Cohorts will be dosed in escalating order, with participants in each cohort (up to n=12 per cohort) randomised in blocks of 4 subjects to receive INI-2004 or placebo at a ratio of 3:1 (active:placebo). INI-2004 or placebo will be administered QW, commencing 2 weeks after administration of the second ragweed nasal allergen challenge.

ELIGIBILITY:
Inclusion Criteria (Phase 1):

1. Participant is willing to refrain from consuming food or beverages containing caffeine and/or xanthene products, within 24 hours prior to check-in on Day -1.
2. Female participants must be of non-child-bearing potential i.e., surgically sterilised at least 6 weeks before the screening visit or postmenopausal.

Inclusion Criteria Phase Ib (Multiple Ascending Dose)

1. Minimum 2 year history of ragweed-induced AR requiring pharmacotherapy (self-reported history accepted) and a positive ragweed skin prick test reaction at Screening Visit.
2. Participant is willing to refrain from consuming food or beverages containing caffeine, within 24 hours prior to each clinic visit.
3. Female participants must be of non-child-bearing potential i.e., surgically sterilised or postmenopausal.

Exclusion Criteria Phase I and Phase Ib (MAD):

1. Hypersensitivity or other clinically significant reaction to the study drug or its active ingredients.
2. Current treatment or use of any prescription medication within 14 days prior to admission to the clinic on Day -1 of active seasonal and perennial allergic rhinitis, non-allergic rhinitis, rhinosinusitis, or asthma. This includes antihistamines, asthma preventers and relievers, nasal decongestants, IN corticosteroids, and immunotherapy or use of over-the-counter medication/vitamins/supplements within 7 days prior to the first dose of study drug. Exceptions include contraception, paracetamol and standard doses of multivitamins.
3. Any clinically relevant structural nasal abnormalities, i.e., nasal septal perforation, nasal polyps, other nasal malformations or history of frequent nosebleeds, upper respiratory tract infection within 2 weeks prior to screening or first dose administration.
4. History of recurrent migraine headaches within 4 weeks prior to screening.
5. Positive alcohol breath, urine test, HBsAg, HepC virus antibody, or HIV antibody tests.
6. Participant has donated blood or blood products within 3 months prior to first dose administration.
7. Use of tobacco products or nicotine-containing products (including smoking cessation aids such as gum or patches.
8. Participant plans to travel to an area with known environmental ragweed exposures at any time during study participation.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and relationship of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and TEAEs leading to discontinuation of study treatment after a single ascending Dose (SAD) | Baseline, Day 1 then daily through to Day 7 End of Study Visit
  Graded using 5-point scale
Incidence, severity and relationship of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and TEAEs leading to discontinuation of study treatment after multiple ascending doses (MAD) | Baseline = Day 0, Day 14, 21, 28, 35 through to Day 58 End of Study Visit
  Graded using 5-point scale
Number of Participants with a Change from baseline in Vital signs measurements after a single ascending Dose (SAD) | Baseline, Day 1 through to Day 7 End of Study Visit
  Pulse rate [PR], systolic and diastolic blood pressure [BP], temperature, respiratory rate.[RR] and oxygen saturation. Blood pressure will be measured using a sphygmomanometer, body temperature will be measured using a thermometer, Heart rate (HR) is measured using vital sign machine, respiratory rate is measured manually via 60-second count and oxygen saturation is measured using a Oximeter. All abnormal assessments measured as Clinically significant post dose will be recorded as AEs.
Number of Participants with a Change from baseline in Vital signs measurements after multiple ascending doses (MAD) | Baseline = Day 0 through to Day 58 End of Study Visit
  Pulse rate [PR], systolic and diastolic blood pressure [BP], temperature, respiratory rate.[RR] and oxygen saturation. Blood pressure will be measured using a sphygmomanometer, body temperature will be measured using a thermometer, Heart rate (HR) is measured using vital sign machine,respiratory rate is measured manually via 60-second count.[RR] and oxygen saturation is measured using a Oximeter. All abnormal assessments measured as Clinically significant post dose will be recorded as AEs.
Change from baseline in 12-lead electrocardiogram parameters after a single ascending Dose (SAD) | Baseline, Day 1 through to Day 7 End of Study Visit
  12-lead ECGs parameters include but not limited to the measurements of ventricular HR, PR interval, RR interval, QRS duration, QT interval and QTcF. At each protocol scheduled timepoint, ECGs will be performed in triplicate with each replicate separated by at least 1 minute and the full set of triplicates completed within 5 minutes.All Clinically Significant findings post-dose will be recorded as AEs.
Change from baseline in 12-lead electrocardiogram parameters after multiple ascending doses (MAD) | Baseline = Day 0 through to Day 58 End of Study Visit
  12-lead ECGs parameters include but not limited to the measurements of ventricular HR, PR interval, RR interval, QRS duration, QT interval and QTcF. At each protocol scheduled timepoint, ECGs will be performed in triplicate with each replicate separated by at least 1 minute and the full set of triplicates completed within 5 minutes.All Clinically Significant findings post-dose will be recorded as AEs.
Number of Participants with a Change from baseline in Clinical laboratory results after a single ascending Dose (SAD) | Baseline, Day 2 through to Day 7 End of Study Visit
  Hematology - Blood samples will be collected. All safety laboratory assessments will be assessed by a certified local laboratory, using that laboratory's normal ranges. Any clinically significant changes will be recorded as Adverse events. The severity of each AE and SAE will be graded using a 5-point scale
Number of Participants with a Change from baseline in Clinical laboratory results after a single ascending Dose (SAD) | Baseline, Day 2 through to Day 7 End of Study Visit
  Serum chemistry- Blood samples will be collected. All safety laboratory assessments will be assessed by a certified local laboratory, using that laboratory's normal ranges. Any clinically significant changes will be recorded as Adverse event. The severity of each AE and SAE will be graded using a 5-point scale
Number of Participants with a Change from baseline in Clinical laboratory results after a single ascending Dose (SAD) | Baseline, Day 2 through to Day 7 End of Study Visit
  Urinalysis- Urine samples will be collected. All safety laboratory assessments will be assessed by a certified local laboratory, using that laboratory's normal ranges. Any clinically significant changes will be recorded as Adverse event. The severity of each AE and SAE will be graded using a 5-point scale
Number of Participants with a Change from baseline in Clinical laboratory results after multiple ascending doses (MAD) | Baseline = Day 0, Day 14 and Day 58 End of Study Visit
  Hematology - Blood samples will be collected. All safety laboratory assessments will be assessed by a certified local laboratory, using that laboratory's normal ranges. Any clinically significant changes will be recorded as Adverse event. The severity of each AE and SAE will be graded using a 5-point scale
Number of Participants with a Change from baseline in Clinical laboratory results after multiple ascending doses (MAD) | Baseline = Day 0, Day 14 and Day 58 End of Study Visit
  Serum chemistry- Blood samples will be collected. All safety laboratory assessments will be assessed by a certified local laboratory, using that laboratory's normal ranges. Any clinically significant changes will be recorded as Adverse event. The severity of each AE and SAE will be graded using a 5-point scale
Number of Participants with a Change from baseline in Clinical laboratory results after multiple ascending doses (MAD) | Baseline = Day 0, Day 14 and Day 58 End of Study Visit
  Urinalysis- Urine samples will be collected. All safety laboratory assessments will be assessed by a certified local laboratory, using that laboratory's normal ranges. Any clinically significant changes will be recorded as Adverse event. The severity of each AE and SAE will be graded using a 5-point scale
Change from baseline in Nasal symptoms after a single ascending Dose (SAD) | Baseline, Day 1 through to Day 7 End of Study Visit
  Presence of itching, discomfort, rhinorrhoea, congestion and sneezing are assessed using a 10 cm visual analogue scale [VAS]. The participant will mark on the VAS where they rank their symptoms ranging from "no symptoms" to "worst symptoms ever experienced".
Change from baseline in Nasal symptoms after multiple ascending doses (MAD) | Baseline = Day 0 through to Day 58 End of Study Visit
  Presence of itching, discomfort, rhinorrhoea, congestion and sneezing are assessed individually as a Total Nasal Symptoms Score (TNSS) at different time points pre and post-ragweed allergen challenge in the MAD portion of the study. TNSS is the sum of symptoms scores for nasal congestion, rhinorrhoea, nasal itching, and sneezing (each scored on a scale of 0 to 3 (below) with total possible score of 0 to 12. The criterion used to score each symptom is described below:
  0 = none: no symptoms
  1. = mild
  2. = moderate
  3. = severe
Change from baseline in Nasal irritancy after a single ascending Dose (SAD) | Baseline, Day 1 through to Day 7 End of Study Visit
  Nasal examination
Change from baseline in Nasal irritancy after multiple ascending doses (MAD) | Baseline = Day 0 through to Day 58 End of Study Visit
  Nasal examination
Change from baseline in Spirometry after a single ascending Dose (SAD) | Baseline, Day 1 through to Day 7 End of Study Visit
  Peak expiratory flow [PEF]-Pulmonary function will be assessed using a handheld spirometer at the time points indicated. A minimum of 3 readings should be completed and recorded at each time point. Observed values and changes from baseline for PEF will be summarised at each scheduled time point using descriptive statistics. Unit of measurement used for PEF is l/min.
Change from baseline in Spirometry after a single ascending Dose (SAD) | Baseline, Day 1 through to Day 7 End of Study Visit
  Forced expiratory volume in 1 second [FEV1]- Pulmonary function will be assessed using a handheld spirometer at the time points indicated. A minimum of 3 readings should be completed and recorded at each time point. Observed values and changes from baseline for FEV1 will be summarised at each scheduled time point using descriptive statistics. Unit of measurement used for FEV1 is liters.
Change from baseline in Spirometry after a single ascending Dose (SAD) | Baseline, Day 1 through to Day 7 End of Study Visit
  Forced vital capacity [FVC]- Pulmonary function will be assessed using a handheld spirometer at the time points indicated. A minimum of 3 readings should be completed and recorded at each time point. Observed values and changes from baseline for FVC will be summarised at each scheduled time point using descriptive statistics. Units of measurement used for FVC is liters.
Change from baseline in Spirometry after a single ascending Dose (SAD) | Baseline, Day 1 through to Day 7 End of Study Visit
  Forced expiratory flow over the middle one-half of the FVC [FEF25-75%]- Pulmonary function will be assessed using a handheld spirometer at the time points indicated. A minimum of 3 readings should be completed and recorded at each time point. Observed values and changes from baseline for spirometry assessments FEF25-75% will be summarised at each scheduled time point using descriptive statistics. Unit of measurement used for FEV1/FVC is %.
Change from baseline in Spirometry after a single ascending Dose (SAD) | Baseline, Day 1 through to Day 7 End of Study Visit
  FEV1/FVC ratio- Pulmonary function will be assessed using a handheld spirometer at the time points indicated. A minimum of 3 readings should be completed and recorded at each time point. Observed values and changes from baseline for spirometry assessments FEV1/FVC ratio will be summarised at each scheduled time point using descriptive statistics. Unit of measurement used for FEF 25%-75% is l/s.
Change from baseline in Spirometry after multiple ascending doses (MAD) | Baseline = Day 0 through to Day 58 End of Study Visit
  Peak expiratory flow [PEF]- Pulmonary function will be assessed using a handheld spirometer at the time points indicated. A minimum of 3 readings should be completed and recorded at each time point. Observed values and changes from baseline for PEF will be summarised at each scheduled time point using descriptive statistics. Unit of measurement used for PEF is l/min.
Change from baseline in Spirometry after multiple ascending doses (MAD) | Baseline = Day 0 through to Day 58 End of Study Visit
  Forced expiratory volume in 1 second [FEV1]- Pulmonary function will be assessed using a handheld spirometer at the time points indicated. A minimum of 3 readings should be completed and recorded at each time point. Observed values and changes from baseline for FEV1 will be summarised at each scheduled time point using descriptive statistics. Unit of measurement used for FEV1 is liters.
Change from baseline in Spirometry after multiple ascending doses (MAD) | Baseline = Day 0 through to Day 58 End of Study Visit
  Forced vital capacity [FVC]- Pulmonary function will be assessed using a handheld spirometer at the time points indicated. A minimum of 3 readings should be completed and recorded at each time point. Observed values and changes from baseline for FVC will be summarised at each scheduled time point using descriptive statistics. Units of measurement used for FVC is liters.
Change from baseline in Spirometry after multiple ascending doses (MAD) | Baseline = Day 0 through to Day 58 End of Study Visit
  FEF25-75% - Pulmonary function will be assessed using a handheld spirometer at the time points indicated. A minimum of 3 readings should be completed and recorded at each time point. Observed values and changes from baseline for FEF25-75%, will be summarised at each scheduled time point using descriptive statistics. Unit of measurement used for FEV1/FVC is %.
Change from baseline in Spirometry after multiple ascending doses (MAD) | Baseline = Day 0 through to Day 58 End of Study Visit
  FEV1/FVC ratio- Pulmonary function will be assessed using a handheld spirometer at the time points indicated. A minimum of 3 readings should be completed and recorded at each time point. Observed values and changes from baseline for FEV1/FVC ratio will be summarised at each scheduled time point using descriptive statistics. Unit of measurement used for FEF 25%-75% is l/s.

SECONDARY OUTCOMES:
Effectiveness of INI-2004 on nasal congestion will be assessed by response to the ragweed allergen challenge (Phase Ib [MAD] only) on Days 14, 21, 23, 28, 35, 37, 51 and 58 compared to baseline (Day 0) | Baseline = Day 0 through to Day 58
  Determined by acoustic rhinometry. Acoustic rhinometry will be performed using GM Instruments. Measurements to include (at a minimum) nasal volume and cross-sectional area. Measurements will be performed for both left and right nasal cavities independently.
Effectiveness of INI-2004 on peak nasal inspiratory flow will be assessed by response to the ragweed allergen challenge (Phase Ib [MAD] only) on Days 14, 21, 23, 28, 35, 37, 51 and 58 compared to baseline (Day 0) | Baseline = Day 0 through to Day 58
  Peak nasal inspiratory flow to be determined using the mean of three replicates.
Effectiveness of INI-2004 on nasal symptoms will be assessed by response to the ragweed allergen challenge (Phase Ib [MAD] only) on Days 23, 37, 51 and 58 compared to baseline (Day 0) | Baseline = Day 0 through to Day 58
  Total nasal symptom score [TNSS] will be measured on a scale of 0 to 3 with a total possible score of 0 to 12. 0= none, no symptoms, 1= mild, 2= moderate, 3=severe.
Effectiveness of INI-2004 on nasal irritancy will be assessed by response to the ragweed allergen challenge (Phase Ib [MAD] only) on Days 23, 37, 51 and 58 compared to baseline (Day 0) | Baseline = Day 0 through to Day 58 End of Study Visit
  Nasal examination- A macroscopic nasal examination will be performed, including conventional anterior rhinoscopy using an otoscope with an attached otic speculum (or nasal speculum and headlight) to assess swelling of the mucosa, erythema, and secretions. All post-dose CS events will be recorded as AEs.
The effectiveness of INI-2004 on Spirometry will be assessed by response to the ragweed allergen challenge (Phase Ib [MAD] only) on Days 23, 37, 51, and 58 compared to baseline (Day 0) via PEF | Baseline = Day 0 through to Day 58
  PEF- Unit of measurement or PEFis l/min
The effectiveness of INI-2004 on Spirometry will be assessed by response to the ragweed allergen challenge (Phase Ib [MAD] only) on Days 23, 37, 51 and 58 compared to baseline (Day 0) Via FEV1 | Baseline = Day 0 through to Day 58
  FEV1- FEV1 is measured in liters
The effectiveness of INI-2004 on Spirometry will be assessed by response to the ragweed allergen challenge (Phase Ib [MAD] only) on Days 23, 37, 51 and 58 compared to baseline (Day 0) via FVC | Baseline = Day 0 through to Day 58
  FVC is measured in liters
The effectiveness of INI-2004 on Spirometry will be assessed by response to the ragweed allergen challenge (Phase Ib [MAD] only) on Days 23, 37, 51 and 58 compared to baseline (Day 0) via FEV1/FVC ratio | Baseline = Day 0 through to Day 58
  FEV1/FVC- is measured in %
The effectiveness of INI-2004 on Spirometry will be assessed by response to the ragweed allergen challenge (Phase Ib [MAD] only) on Days 23, 37, 51 and 58 compared to baseline (Day 0) via FEF | Baseline = Day 0 through to Day 58
  FEF 25%-75%- is measured as l/s
Single dose PK parameters: maximum observed concentration (Cmax) | Day 1 pre dose, then at 15 and 30 mins post-dose, then 1, 2 and 4 hours post-dose, Day 2 at 24 hours post-dose.
  Pharmacokinetics (PK) of INI-2004 in blood plasma following single dose
Single dose PK parameters: Time to Cmax (Tmax) | Day 1 pre dose, then at 15 and 30 mins post-dose, then 1, 2 and 4 hours post-dose, Day 2 at 24 hours post-dose.
  Pharmacokinetics (PK) of INI-2004 in blood plasma following single dose
Single dose PK parameters: Area under the concentration-time curve from time 0 to time t (AUC0-t) | Day 1 pre dose, then at 15 and 30 mins post-dose, then 1, 2 and 4 hours post-dose, Day 2 at 24 hours post-dose.
  Pharmacokinetics (PK) of INI-2004 in blood plasma following single dose
Single dose PK parameters: Area under the concentration-time curve from time 0 to the last measurable concentration (AUClast) | Day 1 pre dose, then at 15 and 30 mins post-dose, then 1, 2 and 4 hours post-dose, Day 2 at 24 hours post-dose.
  Pharmacokinetics (PK) of INI-2004 in blood plasma following single dose
Single dose PK parameters: Half-life (t1/2) | Day 1 pre dose, then at 15 and 30 mins post-dose, then 1, 2 and 4 hours post-dose, Day 2 at 24 hours post-dose.
  Pharmacokinetics (PK) of INI-2004 in blood plasma following single dose
Single dose PK parameters: Clearance (Cl/f) | Day 1 pre dose, then at 15 and 30 mins post-dose, then 1, 2 and 4 hours post-dose, Day 2 at 24 hours post-dose.
  Pharmacokinetics (PK) of INI-2004 in blood plasma following single dose
Single dose PK parameters: Volume of distribution (Vz/f) | Day 1 pre dose, then at 15 and 30 mins post-dose, then 1, 2 and 4 hours post-dose, Day 2 at 24 hours post-dose.
  Pharmacokinetics (PK) of INI-2004 in blood plasma following single dose
Single dose PK parameters: Area under the drug concentration-time curve from time zero infinity (AUCinf) | Day 1 pre dose, then at 15 and 30 mins post-dose, then 1, 2 and 4 hours post-dose, Day 2 at 24 hours post-dose.
  Pharmacokinetics (PK) of INI-2004 in blood plasma following single dose
Multiple dose PK parameters: Drug concentrations from pre-dose to 4 hours post-dose on Days 14 and 35. | Day 14 pre dose then 1, 2 and 4 hours post-dose, Day 35 pre dose then 1, 2 and 4 hours post-dose
  Pharmacokinetics (PK) of INI-2004 in blood plasma following multiple doses
Multiple dose PK parameters: AUC0-4 on Days 14 and 35 (if data permits) | Day 14 pre dose then 1, 2 and 4 hours post-dose, Day 35 pre dose then 1, 2 and 4 hours post-dose
  Pharmacokinetics (PK) of INI-2004 in blood plasma following multiple doses
Multiple dose PK parameters: Post-dose urine drug concentration on Day 14. | Urine to be collected at 0-2 hours post-dose interval on Day 14 only.
  Pharmacokinetics (PK) of INI-2004 in urine following multiple doses - decision if endpoint will be evaluated will be determined following review of plasma PK data from Phase I (SAD).
Single dose PD parameters: Changes in cytokine levels in nasal secretions post-dose compared to baseline pre-dose. | Baseline Day 1 pre-dose then 4, 24 and 48 hours post-dose.
  Pharmacodynamics (PD) of INI-2004 in nasal secretions following single dose
Single dose PD parameters: Changes in cytokine levels in plasma post-dose compared to baseline pre-dose. | Baseline Day 1 pre-dose then 4, 24 and 48 hours post-dose.
  Pharmacodynamics (PD) of INI-2004 in blood plasma following single dose
Multiple dose PD parameters: Changes in concentrations of pro-inflammatory cytokines and nasal mediators in nasal secretions following dose administration compared to baseline pre-dose. | Baseline pre-dose on Day 14 and 35, post-dose Days 14 and 35.
  Pharmacodynamics (PD) of INI-2004 in nasal secretions following multiple doses
Multiple dose PD parameters: Changes in concentrations of pro-inflammatory cytokines and nasal mediators in plasma following dose administration compared to baseline pre-dose. | Baseline pre-dose on Day 14 and 35, post-dose Days 14 and 35.
  Pharmacodynamics (PD) of INI-2004 in blood plasma following multiple doses

OTHER OUTCOMES:
Multiple dose PD parameters: Changes from baseline of IgG | Day 51 pre ragweed challenge.
  Effects of INI-2004 in blood serum on ragweed-specific immunoglobulins following multiple doses.
Multiple dose PD parameters: Changes from baseline of IgE | Day 51 pre ragweed challenge.
  Effects of INI-2004 in blood serum on ragweed-specific immunoglobulins following multiple
Multiple dose PD parameters: Changes from baseline of IgE/IgG | Day 51 pre ragweed challenge.
  Effects of INI-2004 in blood serum on ragweed-specific immunoglobulins following multiple

CONTACTS AND LOCATIONS:
Overall Officials: JonL. Ruckle, Study Director — Inimmune Corp
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No